CLINICAL TRIAL: NCT06078241
Title: Intravenous Lidocaine Infusion Versus Ultrasound Guided Erector Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Postoperative Analgesia in Patients Undergoing Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 556/ 2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous lidocaine infusion (Active Comparator)
  Interventions: Drug: Intravenous lidocaine infusion
- Erector spinae plane block (ESPB) (Active Comparator)
  Interventions: Other: Erector spinae plane block (ESPB)
- Intravenous infusion of normal saline and ESPB with normal saline (Placebo Comparator)
  Interventions: Other: Intravenous infusion of normal saline; Other: ESPB with normal saline

INTERVENTIONS:
Drug: Intravenous lidocaine infusion — Intravenous lidocaine infusion
  Arms: Intravenous lidocaine infusion
Other: Erector spinae plane block (ESPB) — Unilateral erector spinae plane block
  Arms: Erector spinae plane block (ESPB)
Other: Intravenous infusion of normal saline — Intravenous infusion of normal saline
  Arms: Intravenous infusion of normal saline and ESPB with normal saline
Other: ESPB with normal saline — Unilateral ESPB with normal saline
  Arms: Intravenous infusion of normal saline and ESPB with normal saline

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is a minimally invasive procedure to remove stones from the kidney by a small puncture wound through the skin. Patients receiving lidocaine infusion had lower pain scores, reduced postoperative analgesic requirements and decreased intraoperative anesthetic requirements. Erector spinae plane block (ESPB) seems to be effective when compared with no block or a placebo block.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) score I-II..
* Body mass index < 35 kg/m2.

Exclusion Criteria:

* Patient's refusal.
* Known coagulopathy.
* Known peripheral neuropathy or neurological deficits.
* Chronic pain disorders.
* Known allergy to study drugs

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 24 hours postoperatively
  Time to first rescue analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No